CLINICAL TRIAL: NCT01344057
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated, Adjuvanted With MF59C.1 Influenza Vaccine, Formulation 2011-2012, When Administered to Elderly Subjects
Brief Title: Study to Evaluate Safety and Immunogenicity of Sub-unit Adjuvanted Influenza Vaccine Administered to Elderly Subjects, Formulation 2011-2012
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70_32S; 2010-021841-38 (EudraCT Number)
Record Dates: First submitted 2011-04-21; First posted 2011-04-28 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Seasonal Influenza
Keywords: Seasonal Influenza, vaccine

ARMS (1):
- Sub unit, Inactivated, MF59C.1 Adjuvanted Influenza Vaccine (Other): No comparator is administered, only one IM single dose of trivalent subunit inactivated influenza vaccine is administered during the vaccination visit
  Interventions: Biological: Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Seasonal Influenza Vaccine — This phase II is performed as a multicenter study in elderly subjects. Enrolled subjects received one single IM dose of trivalent subunit inactivated adjuvanted flu vaccine during the vaccination visit, according to the study protocol (follow-up period: until day 22) .

SUMMARY:
This study will evaluate the safety and immunogenicity of a sub-unit, adjuvanted Influenza Vaccine Administered to Elderly Subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females volunteers of 65 years of age or older, mentally competent, willing and able to give written informed consent prior to study entry.
* Individuals able to comply with all the study requirements.
* Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.
* Written informed consent must be obtained for all the subjects before enrollment into the study after the nature of the study has been explained.

Key Exclusion Criteria:

* Individuals with any serious chronic or acute disease.
* Individuals with history of any anaphylactic reaction and/or serious allergic reaction following a vaccination.
* Individuals with known or suspected impairment/alteration of immune function.
* Individuals with known or suspected history of drug or alcohol abuse.
* Individuals with a bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject.
* Individuals within the past 6 months, they have: had any seasonal or pandemic laboratory confirmed influenza disease; received any seasonal or pandemic influenza vaccine.
* Individuals with any acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the last 7 days.
* Individuals that have experienced fever (i.e., axillary temperature ≥38°C) within the last 3 days of intended study vaccination.
* Individuals participating in any clinical trial with another investigational product 4 weeks prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
* Individuals who received any other vaccines within 4 weeks prior to enrollment in this study or who are planning to receive any vaccine within 4 weeks from the study vaccines.
* Individuals who are part of study personnel or close family members conducting this study.
* BMI > 35 kg/m2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G. D'Annunzio, Via Dei Vestini, Chieti
  - Department of "Scienze della Salute" University of Genova Via Pastore 1, Genova
  - Satellite: "ASL Lanciano - Vasto", sede legale Via S Spaventa 37, Lanciano
  - Satellite: "Distretto Sanitario di Base di Fossacesia" in Via Polidoro-Vasto, Lanciano
  - Vaccine and Immunotherapy Research Center Department of Infectious and Tropical Diseases San Raffaele Scientific Institute Via Stamira d'Ancona 20, Milan
  - Department of "malattie infettive" Ospedale San Gerardo, via Pergolesi 33, Monza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 63 participants were ≥65 years of age were enrolled at 4 sites in Italy.
Pre-assignment Details: Blood sample for immunogenicity assays were collected before vaccination (Day 1) and after 21 Days.
Groups:
- FLUAD: Participants received a single intramuscular (IM) dose of 0.5 milliliter (mL) of FLUAD containing 15μg each of the three influenza antigens into the deltoid region of the non-dominant arm during the vaccination visit, according to the study protocol until day 22.
Period: Overall Study
Arm/Group | FLUAD
Started | 63
Completed | 62
Not Completed | 1
Not completed — Premature Withdrawal | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was defined as all participants who were enrolled into the study.
Groups:
- FLUAD: Participants received a single IM dose of 0.5 mL of FLUAD containing 15μg each of the three influenza antigens into the deltoid region of the non-dominant arm during the vaccination visit, according to the study protocol until day 22.
Arm/Group | FLUAD
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Seroconversion or Significant Increase in Single Radial Hemolysis (SRH) Area Against Each of Three Vaccine Strains After One Vaccination of FLUAD
Description: Immunogenicity was measured as the percentage of participants who achieved seroconversion or significant increase in single radial hemolysis (SRH) area, against each of the three vaccine strains, three weeks after vaccination (day 22), evaluated using SRH assay.
  Seroconversion: proportion of participants with negative pre-vaccination serum and a post-vaccination serum area ≥ 25 mm2. Significant increase: proportion of participants with at least a 50% increase in area from positive pre-vaccination serum. Seroconversion or significant increase: proportion of participants with either seroconversion or significant increase.
  The European (Committee for Medicinal Products for Human Use [CHMP]) criterion is met, if percentage of participants achieving seroconversion or significant increase in SRH area is 30% (≥65 years).
Time Frame: day 22
Population: Per protocol (PP) analysis set included all enrolled participants who had correctly received the vaccine, provided evaluable serum samples before and after vaccination, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLUAD
Number analyzed (Participants) | 63
Percentage of participants
  A/H1N1 (N= 62) | 69 [56 to 80]
  A/H3N2 (N= 62) | 50 [37 to 63]
  B (N= 62) | 26 [16 to 38]

2. Secondary Outcome: Number of Participants Who Reported Solicited Local and Systemic Reactions
Description: Safety was assessed for participants who reported solicited local and systemic reactions from day 1 up to and including day 4 after the FLUAD vaccination.
Time Frame: 1 to 4 days post-vaccination
Population: Analysis was done using the safety dataset; participants who received study vaccination and who provided post-vaccination safety data.
Measure: Number; unit: Number of participants
Arm/Group | FLUAD
Number analyzed (Participants) | 63
Number of participants
  Injection site ecchymosis (N= 62) | 3
  Injection site erythema (N= 62) | 7
  Injection site induration (N= 62) | 4
  Injection site swelling (N= 62) | 7
  Injection site pain (N= 62) | 21
  Chills Shivering (N= 62) | 4
  Malaise (N= 62) | 3
  Myalgia (N= 62) | 6
  Arthralgia (N= 62) | 4
  Headache (N= 62) | 4
  Sweating (N= 62) | 1
  Fatigue (N= 62) | 2
  Fever (≥38°C) (N= 61) | 0

3. Primary Outcome: Geometric Mean Ratio of Participants Against Each of the Three Vaccine Strains After One Vaccination of FLUAD
Description: Geometric mean ratio (GMR) of participants was calculated as the ratio of post-vaccination to pre-vaccination SRH geometric mean areas (GMAs), directed against each of the three vaccine strains, three weeks after FLUAD vaccination (day 22).
  The CHMP criterion was met if the geometric mean increase (GMR, day 22/day 1) in SRH antibody area is >2.0 (≥65 years).
Time Frame: day 22
Population: Analysis was done using PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | FLUAD
Number analyzed (Participants) | 63
Ratio
  A/H1N1 (N= 62) | 2.54 [2.1 to 3.07]
  A/H3N2 (N= 62) | 1.9 [1.63 to 2.2]
  B (N= 62) | 1.36 [1.21 to 1.53]

4. Primary Outcome: Percentage of Participants Who Achieved SRH Area ≥25mm2 Against Each of the Three Vaccine Strains After One Vaccination of FLUAD
Description: Immunogenicity was measured as the percentage of participants achieving SRH area ≥25 mm2 against each of the three vaccine strains at baseline (day 1) and three weeks after FLUAD vaccination (day 22).
  This criterion is met according to CHMP guideline if percentage of participants achieving SRH area ≥25 mm2 is 60% (≥65 years).
Time Frame: day 22
Population: Analysis was done using PP set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLUAD
Number analyzed (Participants) | 63
Percentage of participants
  A/H1N1 (N= 62) | 89 [78 to 95]
  A/H3N2 (N= 62) | 69 [56 to 80]
  B (N= 62) | 94 [84 to 98]

ADVERSE EVENTS:
Time Frame: From Day 1 through Day 22.
Description: Adverse events other than local and systemic reactions or solicited reactions lasting longer than 3 days after vaccination were documented during the study period.
Groups:
- FLUAD: Participants received a single IM 0.5 mL dose of trivalent subunit inactivated adjuvanted influenza vaccine FLUAD during the vaccination visit, according to the study protocol (follow-up period: until day 22).
Arm/Group | FLUAD
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 6/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLUAD (N=63)
Injection site erythema (General disorders) | 3
Injection site haemorrhage (General disorders) | 2
Injection site induration (General disorders) | 2
Injection site pain (General disorders) | 2
Injection site swelling (General disorders) | 2
Mastoiditis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.